CLINICAL TRIAL: NCT02586415
Title: Endovascular Therapy Following Imaging Evaluation for Ischemic Stroke 3
Acronym: DEFUSE 3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed a high likelihood of benefit in the endovascular group
Sponsor: Gregory W Albers (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Cincinnati (Other); Medical University of South Carolina (Other); NINDS Stroke Trials Network (StrokeNet) (Other)
Responsible Party: Sponsor-Investigator, Gregory W Albers, Professor of Neurology, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116661; U10NS086487 (NIH); U01NS092076 (NIH)
Record Dates: First submitted 2015-10-21; First posted 2015-10-26 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Stroke, Acute; Cerebral Infarction
Keywords: endovascular; endovascular procedure; Mechanical Thrombectomy
MeSH Terms: conditions — Stroke; Cerebral Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- endovascular thrombectomy therapy (Active Comparator): Treatment with one or more thrombectomy devices (only the devices listed in this protocol are approved for use in DEFUSE 3) plus standard medical therapy for patients who have evidence of an ICA or MCA M1 occlusion and a Target Mismatch Profile.
  Devices approved for use in DEFUSE 3:
  * Trevo Retriever
  * Solitaire™ FR Revascularization Device
  * Penumbra thrombectomy system
  * Covidien MindFrame Capture Revascularization Device
  Interventions: Procedure: Endovascular Thrombectomy; Device: Trevo Retriever; Device: Solitaire™ FR Revascularization Device; Device: Penumbra thrombectomy system; Device: Covidien MindFrame Capture Revascularization Device
- Medical Management (No Intervention): standard medical therapy alone

INTERVENTIONS:
Procedure: Endovascular Thrombectomy — Patients will be treated with thrombectomy devices (stent-retrievers) and/or suction thrombectomy systems currently cleared by the FDA for thrombus removal in patients experiencing an acute stroke following the published instructions for use for these devices. These devices will be used between 6 and 16 hours following symptom onset in DEFUSE 3 based on an FDA IDE. The devices which will be used are the Trevo Retriever, the Solitaire Revascularization Device and the Penumbra system thrombectomy system.
  Arms: endovascular thrombectomy therapy
Device: Trevo Retriever — Trevo Retriever is one of the interventional devices that is approved for use in DEFUSE 3 during the endovascular thrombectomy procedure. The device choice is at the discretion of the physician performing the procedure.
  Arms: endovascular thrombectomy therapy
Device: Solitaire™ FR Revascularization Device — Solitaire™ FR Revascularization Device is one of the interventional devices that is approved for use in DEFUSE 3 during the endovascular thrombectomy procedure. The device choice is at the discretion of the physician performing the procedure.
  Arms: endovascular thrombectomy therapy
Device: Penumbra thrombectomy system — Penumbra thrombectomy system is one of the interventional devices that is approved for use in DEFUSE 3 during the endovascular thrombectomy procedure. The device choice is at the discretion of the physician performing the procedure. The Penumbra System includes:
  • Penumbra Aspiration Pump (1115V) Penumbra System 054 Penumbra System MAX Penumbra System 110 Aspiration Tubing Penumbra System [026, 032, 041] Penumbra System Separator Flex [026, 032, 041, 054] Penumbra Pump MAX Penumbra System Reperfusion Catheter ACE64 & ACE68
  Arms: endovascular thrombectomy therapy
Device: Covidien MindFrame Capture Revascularization Device — Covidien MindFrame Capture Revascularization Device is one of the interventional devices that is approved for use in DEFUSE 3 during the endovascular thrombectomy procedure. The device choice is at the discretion of the physician performing the procedure.
  Arms: endovascular thrombectomy therapy

SUMMARY:
This is a study to evaluate the hypothesis that FDA cleared thrombectomy devices plus medical management leads to superior clinical outcomes in acute ischemic stroke patients at 90 days when compared to medical management alone in appropriately selected subjects with the Target mismatch profile and an MCA (M1 segment) or ICA occlusion who can be randomized and have endovascular treatment initiated between 6-16 hours after last seen well.

DETAILED DESCRIPTION:
DEFUSE 3 is a prospective randomized Phase III multicenter controlled trial of patients with acute ischemic anterior circulation strokes due to large artery occlusion treated between 6-16 hours of stroke onset with endovascular thrombectomy therapy vs. control.

The primary endpoint, the modified Rankin Score, will be assessed at 3 months. The patients' participation in the study concludes at that time (3 months from stroke onset). The study will randomize up to 476 patients over 4 years. The purpose of DEFUSE 3 is to assess the safety and efficacy of thrombectomy in carefully selected patients in an extended time window. Only the devices listed in this protocol will be used. Selection of the specific device (or devices) is determined by the individual endovascular therapist.

Patients who meet the inclusion criteria will undergo either CT Perfusion/CT Angiogram or MR DWI/PWI/MRA studies prior to randomization. Patients who have evidence of an ICA or MCA M1 occlusion and a Target Mismatch Profile will be randomized in a 1:1 ratio to treatment with one or more DEFUSE 3 approved thrombectomy devices (only the devices listed in this protocol are approved for use in DEFUSE 3) plus standard medical therapy versus standard medical therapy alone. Patients who are enrolled, but not randomized, will receive standard therapy according to local guidelines. Baseline data, and information about early stroke therapies, will be captured for this group of patients.

Randomization of a maximum of 476 patients is planned. A novel adaptive design will identify, at interim analyses, the group with the best prospect for showing benefit from endovascular treatment, based on baseline core lesion volumes and the times since stroke onset. Interim analyses will be conducted at 200 and 340 patients, at which time the study may stop for efficacy/futility, or the inclusion criteria may be adjusted in the case of futility.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Signs & symptoms consistent w/ the diagnosis of acute anterior circulation ischemic stroke
2. Age 18-90 years
3. Baseline NIHSSS is ≥ 6 and remains ≥6 immediately prior to randomization
4. Endovascular treatment can be initiated (femoral puncture) between 6 and 16 hours of stroke onset. Stroke onset is defined as the time the patient was last known to be at their neurologic baseline (wake-up strokes are eligible if they meet the above time limits).
5. modified Rankin Scale less than or equal to 2 prior to qualifying stroke (functionally independent for all ADLs)
6. Patient/Legally Authorized Representative has signed the Informed Consent form.

Clinical Exclusion Criteria:

1. Other serious, advanced, or terminal illness (investigator judgment) or life expectancy is less than 6 months.
2. Pre-existing medical, neurological or psychiatric disease that would confound the neurological or functional evaluations
3. Pregnant
4. Unable to undergo a contrast brain perfusion scan with either MRI or CT
5. Known allergy to iodine that precludes an endovascular procedure
6. Treated with tPA >4.5 hours after time last known well
7. Treated with tPA 3-4.5 hours after last known well AND any of the following; age >80, current anticoagulant use, history of diabetes or prior stroke, NIHSS >25
8. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; recent oral anticoagulant therapy with INR > 3 (recent use of one of the new oral anticoagulants is not an exclusion if estimated GFR > 30 ml/min).
9. Seizures at stroke onset if it precludes obtaining an accurate baseline NIHSS
10. Baseline blood glucose of <50mg/dL (2.78 mmol) or >400mg/dL (22.20 mmol)
11. Baseline platelet count < 50,000/uL
12. Severe, sustained hypertension (Systolic BP >185 mmHg or Diastolic BP >110 mmHg)
13. Current participation in another investigational drug or device study
14. Presumed septic embolus; suspicion of bacterial endocarditis
15. Clot retrieval attempted using a neurothrombectomy device prior to 6 hrs from symptom onset
16. Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject if an endovascular procedure was performed.

Neuroimaging Inclusion Criteria:

1. ICA or MCA-M1 occlusion (carotid occlusions can be cervical or intracranial; with or without tandem MCA lesions) by MRA or CTA

   AND
2. Target Mismatch Profile on CT perfusion or MRI (ischemic core volume is < 70 ml, mismatch ratio is >/= 1.8 and mismatch volume* is >/= 15 ml)

Alternative neuroimaging inclusion criteria (if perfusion imaging or CTA/MRA is technically inadequate):

A) If CTA (or MRA) is technically inadequate:

Tmax>6s perfusion deficit consistent with an ICA or MCA-M1 occlusion AND Target Mismatch Profile (ischemic core volume is < 70 ml, mismatch ratio is >1.8 and mismatch volume is >15 ml as determined by RAPID software)

B) If MRP is technically inadequate:

ICA or MCA-M1 occlusion (carotid occlusions can be cervical or intracranial; with or without tandem MCA lesions) by MRA (or CTA, if MRA is technically inadequate and a CTA was performed within 60 minutes prior to the MRI) AND DWI lesion volume < 25 ml

C) If CTP is technically inadequate:

Patient can be screened with MRI and randomized if neuroimaging criteria are met.

Neuroimaging Exclusion Criteria:

1. ASPECTS score <6 on non-contrast CT (if patient is enrolled based on CT perfusion criteria)
2. Evidence of intracranial tumor (except small meningioma) acute intracranial hemorrhage, neoplasm, or arteriovenous malformation
3. Significant mass effect with midline shift
4. Evidence of internal carotid artery dissection that is flow limiting or aortic dissection
5. Intracranial stent implanted in the same vascular territory that precludes the safe deployment/removal of the neurothrombectomy device
6. Acute symptomatic arterial occlusions in more than one vascular territory confirmed on CTA/MRA (e.g., bilateral MCA occlusions, or an MCA and a basilar artery occlusion).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Albers, MD, Principal Investigator — Stanford University; Michael Marks, MD, Principal Investigator — Stanford University; Maarten Lansberg, MD, PhD, Principal Investigator — Stanford University
Locations (40):
- United States (40):
  - University of Alabama, Birmingham, Alabama
  - Community Regional Medical Center, Fresno, California
  - Scripps Memorial Hospital, La Jolla, California
  - UCSD Medical Center/Hillcrest Hospital, La Jolla, California
  - Keck Hospital of University of Southern California, Los Angeles, California
  - UCSF Medical Center, San Francisco, CA, San Francisco, California
  - Stanford University, Stanford, California
  - John Muir Medical Center, Walnut Creek, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - The Valley Hospital, Ridgewood, New Jersey
  - Mount Sinai Hospital, New York, New York
  - New York Presbyterian Hospital at Columbia, New York, New York
  - NYP Weill Cornell Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Health Richland, Columbia, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University Medical Center Brackenridge, Austin, Texas
  - Seton Medical Center/UT Southwestern, Austin, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Utah Healthcare, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Albers GW, Lansberg MG, Kemp S, Tsai JP, Lavori P, Christensen S, Mlynash M, Kim S, Hamilton S, Yeatts SD, Palesch Y, Bammer R, Broderick J, Marks MP. A multicenter randomized controlled trial of endovascular therapy following imaging evaluation for ischemic stroke (DEFUSE 3). Int J Stroke. 2017 Oct;12(8):896-905. doi: 10.1177/1747493017701147. Epub 2017 Mar 24. PMID 28946832
- [Result] Albers GW, Marks MP, Kemp S, Christensen S, Tsai JP, Ortega-Gutierrez S, McTaggart RA, Torbey MT, Kim-Tenser M, Leslie-Mazwi T, Sarraj A, Kasner SE, Ansari SA, Yeatts SD, Hamilton S, Mlynash M, Heit JJ, Zaharchuk G, Kim S, Carrozzella J, Palesch YY, Demchuk AM, Bammer R, Lavori PW, Broderick JP, Lansberg MG; DEFUSE 3 Investigators. Thrombectomy for Stroke at 6 to 16 Hours with Selection by Perfusion Imaging. N Engl J Med. 2018 Feb 22;378(8):708-718. doi: 10.1056/NEJMoa1713973. Epub 2018 Jan 24. PMID 29364767
- [Result] Marks MP, Heit JJ, Lansberg MG, Kemp S, Christensen S, Derdeyn CP, Rasmussen PA, Zaidat OO, Broderick JP, Yeatts SD, Hamilton S, Mlynash M, Albers GW; DEFUSE 3 Investigators. Endovascular Treatment in the DEFUSE 3 Study. Stroke. 2018 Aug;49(8):2000-2003. doi: 10.1161/STROKEAHA.118.022147. PMID 29986935
- [Derived] Yu Y, Christensen S, Ouyang J, Scalzo F, Liebeskind DS, Lansberg MG, Albers GW, Zaharchuk G. Predicting Hypoperfusion Lesion and Target Mismatch in Stroke from Diffusion-weighted MRI Using Deep Learning. Radiology. 2023 Apr;307(1):e220882. doi: 10.1148/radiol.220882. Epub 2022 Dec 6. PMID 36472536
- [Derived] Tate WJ, Polding LC, Christensen S, Mlynash M, Kemp S, Heit JJ, Marks MP, Albers GW, Lansberg MG. Predictors of Early and Late Infarct Growth in DEFUSE 3. Front Neurol. 2021 Jul 1;12:699153. doi: 10.3389/fneur.2021.699153. eCollection 2021. PMID 34276547
- [Derived] Polding LC, Tate WJ, Mlynash M, Marks MP, Heit JJ, Christensen S, Kemp S, Albers GW, Lansberg MG; DEFUSE 3 Investigators. Quality of Life in Physical, Social, and Cognitive Domains Improves With Endovascular Therapy in the DEFUSE 3 Trial. Stroke. 2021 Apr;52(4):1185-1191. doi: 10.1161/STROKEAHA.120.031490. Epub 2021 Feb 18. PMID 33596675
- [Derived] Sarraj A, Mlynash M, Heit J, Pujara D, Lansberg M, Marks M, Albers GW. Clinical Outcomes and Identification of Patients With Persistent Penumbral Profiles Beyond 24 Hours From Last Known Well: Analysis From DEFUSE 3. Stroke. 2021 Mar;52(3):838-849. doi: 10.1161/STROKEAHA.120.031147. Epub 2021 Feb 10. PMID 33563012
- [Derived] Cereda CW, Mlynash M, Cippa PE, Kemp S, Heit JJ, Marks MP, Lansberg MG, Albers GW. Renal Safety of Multimodal Brain Imaging Followed by Endovascular Therapy. Stroke. 2021 Jan;52(1):313-316. doi: 10.1161/STROKEAHA.120.030816. Epub 2020 Nov 30. PMID 33250038
- [Derived] Heit JJ, Mlynash M, Christensen S, Kemp SM, Lansberg MG, Marks MP, Olivot JM, Gregory AW. What predicts poor outcome after successful thrombectomy in late time windows? J Neurointerv Surg. 2021 May;13(5):421-425. doi: 10.1136/neurintsurg-2020-016125. Epub 2020 Jun 17. PMID 32554693
- [Derived] Kim-Tenser M, Mlynash M, Lansberg MG, Tenser M, Bulic S, Jagadeesan B, Christensen S, Simpkins A, Albers GW, Marks MP, Heit JJ. CT perfusion core and ASPECT score prediction of outcomes in DEFUSE 3. Int J Stroke. 2021 Apr;16(3):288-294. doi: 10.1177/1747493020915141. Epub 2020 Mar 31. PMID 32233746
- [Derived] Dula AN, Mlynash M, Zuck ND, Albers GW, Warach SJ; DEFUSE 3 Investigators. Neuroimaging in Ischemic Stroke Is Different Between Men and Women in the DEFUSE 3 Cohort. Stroke. 2020 Feb;51(2):481-488. doi: 10.1161/STROKEAHA.119.028205. Epub 2019 Dec 12. PMID 31826731
- [Derived] Amukotuwa SA, Fischbein NJ, Albers GW, Davis S, Donnan GA, Andre JB, Bammer R. Comparison of T2*GRE and DSC-PWI for hemorrhage detection in acute ischemic stroke patients: Pooled analysis of the EPITHET, DEFUSE 2, and SENSE 3 stroke studies. Int J Stroke. 2020 Feb;15(2):216-225. doi: 10.1177/1747493019858781. Epub 2019 Jul 10. PMID 31291850
- [Derived] Tate WJ, Polding LC, Kemp S, Mlynash M, Heit JJ, Marks MP, Albers GW, Lansberg MG. Thrombectomy Results in Reduced Hospital Stay, More Home-Time, and More Favorable Living Situations in DEFUSE 3. Stroke. 2019 Sep;50(9):2578-2581. doi: 10.1161/STROKEAHA.119.025165. Epub 2019 Jul 10. PMID 31288666
- [Derived] Heit JJ, Mlynash M, Kemp SM, Lansberg MG, Christensen S, Marks MP, Ortega-Gutierrez S, Albers GW. Rapid Neurologic Improvement Predicts Favorable Outcome 90 Days After Thrombectomy in the DEFUSE 3 Study. Stroke. 2019 May;50(5):1172-1177. doi: 10.1161/STROKEAHA.119.024928. PMID 30932783
- [Derived] Christensen S, Mlynash M, Kemp S, Yennu A, Heit JJ, Marks MP, Lansberg MG, Albers GW. Persistent Target Mismatch Profile >24 Hours After Stroke Onset in DEFUSE 3. Stroke. 2019 Mar;50(3):754-757. doi: 10.1161/STROKEAHA.118.023392. PMID 30735466
- [Derived] Sarraj A, Mlynash M, Savitz SI, Heit JJ, Lansberg MG, Marks MP, Albers GW. Outcomes of Thrombectomy in Transferred Patients With Ischemic Stroke in the Late Window: A Subanalysis From the DEFUSE 3 Trial. JAMA Neurol. 2019 Jun 1;76(6):682-689. doi: 10.1001/jamaneurol.2019.0118. PMID 30734042
- [Derived] Rao V, Christensen S, Yennu A, Mlynash M, Zaharchuk G, Heit J, Marks MP, Lansberg MG, Albers GW. Ischemic Core and Hypoperfusion Volumes Correlate With Infarct Size 24 Hours After Randomization in DEFUSE 3. Stroke. 2019 Mar;50(3):626-631. doi: 10.1161/STROKEAHA.118.023177. PMID 30727840
- [Derived] de Havenon A, Mlynash M, Kim-Tenser MA, Lansberg MG, Leslie-Mazwi T, Christensen S, McTaggart RA, Alexander M, Albers G, Broderick J, Marks MP, Heit JJ; DEFUSE 3 Investigators. Results From DEFUSE 3: Good Collaterals Are Associated With Reduced Ischemic Core Growth but Not Neurologic Outcome. Stroke. 2019 Mar;50(3):632-638. doi: 10.1161/STROKEAHA.118.023407. PMID 30726184
- [Derived] Lansberg MG, Mlynash M, Hamilton S, Yeatts SD, Christensen S, Kemp S, Lavori PW, Ortega-Gutierrez S, Broderick J, Heit J, Marks MP, Albers GW; DEFUSE 3 Investigators. Association of Thrombectomy With Stroke Outcomes Among Patient Subgroups: Secondary Analyses of the DEFUSE 3 Randomized Clinical Trial. JAMA Neurol. 2019 Apr 1;76(4):447-453. doi: 10.1001/jamaneurol.2018.4587. PMID 30688974

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2016 through May 2017, a total of 182 patients underwent randomization (92 to the endovascular-therapy group and 90 to the medical-therapy group) at 38 centers in the United States.
Pre-assignment Details: After obtaining written informed consent, participants were randomized if they met all clinical and imaging eligibility requirements and could undergo initiation of endovascular therapy between 6 and 16 hours after the time that they had last been known to be well.
Groups:
- Endovascular Thrombectomy Therapy: Treatment with one or more thrombectomy devices (only the devices listed in this protocol are approved for use in DEFUSE 3) plus standard medical therapy for patients who have evidence of an ICA or MCA M1 occlusion and a Target Mismatch Profile.
  Devices approved for use in DEFUSE 3:
  * Trevo Retriever
  * Solitaire™ FR Revascularization Device
  * Penumbra thrombectomy system
  * Covidien MindFrame Capture Revascularization Device
  Endovascular Thrombectomy: Patients will be treated with thrombectomy devices (stent-retrievers) and/or suction thrombectomy systems currently cleared by the FDA for thrombus removal in patients experiencing an acute stroke following the published instructions for use for these devices. These devices will be used between 6 and 16 hours following symptom onset in DEFUSE 3 based on an FDA IDE. The devices which will be used are the Trevo Retriever, the Solitaire Revascularization Device and the Penumbra system thrombectomy system.
  Trevo Retriever: Trevo R
Period: Overall Study
Arm/Group | Endovascular Thrombectomy Therapy | Medical Management
Started | 92 | 90
24 Hour Assessment | 91 | 90
Day 30 Assessment | 81 | 70
Day 90 Assessment | 78 | 65
Completed | 78 | 65
Not Completed | 14 | 25
Not completed — Death | 13 | 23
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Endovascular Thrombectomy Therapy: Treatment with one or more thrombectomy devices (only the devices listed in this protocol are approved for use in DEFUSE 3) plus standard medical therapy for patients who have evidence of an ICA or MCA M1 occlusion and a Target Mismatch Profile.
  Devices approved for use in DEFUSE 3:
  * Trevo Retriever
  * Solitaire™ FR Revascularization Device
  * Penumbra thrombectomy system
  * Covidien MindFrame Capture Revascularization Device
  Endovascular Thrombectomy: Patients will be treated with thrombectomy devices (stent-retrievers) and/or suction thrombectomy systems currently cleared by the FDA for thrombus removal in patients experiencing an acute stroke following the published instructions for use for these devices. These devices will be used between 6 and 16 hours following symptom onset in DEFUSE 3 based on an FDA IDE. The devices which will be used are the Trevo Retriever, the Solitaire Revascularization Device and the Penumbra system thrombectomy system.
- Total: Total of all reporting groups
Arm/Group | Endovascular Thrombectomy Therapy | Medical Management | Total
Number analyzed (Participants) | 92 | 90 | 182
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [59 to 78.5] | 71 [59 to 80] | 70.5 [59 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 92
  Male | 46 | 44 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 10 | 24
  Not Hispanic or Latino | 77 | 80 | 157
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 78 | 80 | 158
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
NIHSS, continuous [Median (Inter-Quartile Range); unit: units on a scale] — The NIHSS is a clinician-rated, 15-item scale designed to assess the severity of stroke-related neurological deficits: level of consciousness, eye movements, visual fields, facial symmetry, motor strength (arm and leg), coordination, sensation, language (aphasia and dysarthria), and neglect. Each item is rated on a 3-, 4-, or 5-point scale ranging from 0 (normal) to the maximum score (extremely severe symptoms). The total score of the 15 items ranges from 0 to 42, where lower scores indicate less impairment.
  units on a scale | 16 [10 to 20] | 16 [12 to 21] | 16 [11 to 21]

OUTCOME MEASURES:

1. Primary Outcome: The Distribution of Scores on the Modified Rankin Scale (mRS) at Day 90
Description: The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: Day 90
Population: intention to treat
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Endovascular Thrombectomy Therapy | Medical Management
Number analyzed (Participants) | 92 | 90
score on a scale | 3 [1 to 4] | 4 [3 to 6]
Statistical Analysis 1: Comparison: Endovascular Thrombectomy Therapy vs Medical Management; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Criteria to assess superiority was a two-sided P value of <0.05. The study was terminated early because the pre-specified stopping boundary of P <0.0025 was crossed at the first interim analysis (N=182); Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.63 to 4.70]

2. Secondary Outcome: Count of Patients With mRS 0-2 at Day 90 as a Measure of Functional Independence
Description: The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death. 0 - No symptoms.
  * No significant disability. Able to carry out all usual activities, despite some symptoms.
  * Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  * Moderate disability. Requires some help, but able to walk unassisted.
  * Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  * Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  * Dead.
Time Frame: day 90
Population: intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Therapy | Medical Management
Number analyzed (Participants) | 92 | 90
Participants | 41 | 15

3. Other Pre Specified Outcome: Count of Participants With Symptomatic Intracranial Hemorrhage (Primary Safety Outcome)
Description: Defined as NIHSS worsening of 4 or more points associated with brain hemorrhage within 36 hours of randomization
Time Frame: 36 hours
Measure: Count of Participants; unit: Participants
Groups:
- Endovascular Thrombectomy Therapy: Treatment with one or more thrombectomy devices cleared by the FDA for thrombus removal in patients experiencing an acute stroke.
Arm/Group | Endovascular Thrombectomy Therapy | Medical Management
Number analyzed (Participants) | 92 | 90
Participants | 6 | 4

4. Other Pre Specified Outcome: Parenchymal Hematoma Type 2 (Safety Outcome)
Description: PH 2 rates on the 24 hour scan (±6)
Time Frame: 24 (±6) hours
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Infarct Volume (Imaging Outcome)
Description: Infarct volume on diffusion-weighted MRI (or CT if MRI not feasible) at 24 (±6) hours after randomization
Time Frame: 24 (+/- 6) hours
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Lesion Growth (Imaging Outcome)
Description: Lesion growth between the RAPID-identified ischemic core on baseline imaging and the infarct volume at 24 hours (±6)
Time Frame: 24 hours (±6)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Reperfusion (Imaging Outcome)
Description: Successful reperfusion defined as a >90% reduction in Tmax>6sec lesion volume between baseline and 24 hours
Time Frame: between baseline and 24 hours (+/- 6 hours)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Recanalization (Imaging Outcome)
Description: Recanalization of the primary arterial occlusive lesion at 24-hours on CTA/MRA
Time Frame: 24 hours (±6)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Endovascular Thrombectomy Therapy | Medical Management
All-Cause Mortality (participants affected / at risk) | 13/92 | 23/90
Serious Adverse Events (participants affected / at risk) | 40/92 | 48/90
Other Adverse Events (participants affected / at risk) | 57/92 | 59/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Thrombectomy Therapy (N=92) | Medical Management (N=90)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 4 (4) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery dissection (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 5 (5)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 2 (2)
Haemorrhagic transformation stroke (Nervous system disorders) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 2 (2) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 3 (3) | 9 (9)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Thrombectomy Therapy (N=92) | Medical Management (N=90)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 5 (5)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 4 (4) | 4 (4)
Cerebral infarction (Nervous system disorders) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 5 (5) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 15 (16) | 10 (10)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 5 (5) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 0 (0) | 5 (5)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord oedema (Nervous system disorders) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tenderness (General disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Troponin (Investigations) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 3 (3) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 10 (10)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Vessel perforation (Vascular disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT02586415/SAP_000.pdf
  • Study Protocol (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT02586415/Prot_001.pdf